CLINICAL TRIAL: NCT04659694
Title: The Physical and Psychosocial Effects of a Whole Systems Wellness Intervention for Older Adults Living in Care Homes: A Feasibility Study
Brief Title: Effect of an Intervention on Health in Older Care Home Residents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of PhD
Sponsor: Bournemouth University (Other)
Collaborators: Oomph! Wellness (Unknown); Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government); Solent University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 276089
Record Dates: First submitted 2020-05-21; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Sedentary Behavior; Frail Elderly Syndrome; Frailty; Lifestyle, Sedentary; Life Style Induced Illness
Keywords: elderly; older adults; physical activity; psychosocial activity; care home; care home staff; care home residents
MeSH Terms: conditions — Sedentary Behavior; Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: A mixed method design is an integrative methodology in understanding the social inquiry into the implementation of an intervention(Greene,2008). The whole system wellness intervention will be applied to care home residents by (intervention-trained) care home staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): This study only contains one arm
  Interventions: Other: Wellness programme provided by Oomph! Wellness company

INTERVENTIONS:
Other: Wellness programme provided by Oomph! Wellness company — The Oomph! wellness programme empowers older adults to lead a full life for life. It focuses on building an individual-centred programme that consists of a varied exercise and activity plans including days out. All of these, aims in improving the physical and psychosocial wellness in older adults. This intervention is a three day training session for care home staff to understand and learn how to facilitate care activities within their care home.
  Other Names: Oomph! Wellness

SUMMARY:
Care home residents spent 79% of their time being sedentary. Reduced physical activity and lack of mental stimulation causes general weakness and frailty in older adults that can result in increased healthcare needs. It is important that care home residents spend their time being both physically and psychosocially engaged.

This study aims to investigate the effect of a wellness programme on physical and psychosocial wellbeing in older adults living in care homes. Through this process this study will assess the feasibility of implementing the programme and collecting data in care home settings.

There are two main groups of participants, 1) care home residents and 2) care home staff.

Care home residents will have data collected at three time points. The first time point will be before the intervention (baseline) in the care home setting. The second time point will be three months after the intervention has been delivered. The third time point will be 6 months after the intervention has been delivered.

The following measurements will be conducted:

1. Measuring hand grip strength by having to grip a device as firmly as possible and measurements will be taken,
2. Answering questionnaires about quality of life, daily routine, appetite, thoughts about wellness activities the participants have participated in,
3. Wearing a little 'match box-like' device (that measures daily movements and sleep patterns) for 7 consecutive days.

Care home staff will be invited to participate in a focus group discussion 6 months after the intervention. Hence, this research will aim to understand the impact of a wellness programme that incorporates physical and psychosocial components that targets the holistic wellbeing of older adults.

DETAILED DESCRIPTION:
The following potential issues have been identified:

1. This feasibility study is being carried out in older adults living in care homes. Older adults are considered to be vulnerable population by the definition of the World Health Organisation.
2. This study involves residents with cognitive impairment who may not be able to give consent for themselves to take part in the study. To overcome these issues, the research team is very mindful not to exclude residents with cognitive impairment who otherwise are able to participate in the Wellness activities. Th investigators will strictly adopt the Dewing process of gaining consent for older adults with cognitive impairment which involves ongoing consent monitoring. The investigators have followed the guidelines of Mental Capacity Act 2005 and designed participant information sheets and consulted declaration form who could consent on the participant's behalf (consultee). If consent is not obtained, the participant will not be recruited into the study. The consultee will be able to withdraw consent at any time in the study. Any visible distress observed during participation (eg. use of handgrip dynamometer & accelerometer) will be recorded and the participant will be withdrawn from the study.

   Participants will also be regularly reminded that they can choose to withdraw from the study at any point, without any explanation and that care received would not be affected or compromised due to this study.
3. All data collected will be stored on password protected computers and/or the BU secure server and will be handled in accordance with the General Data Protection Regulation 2018 and Data Protection Act 2018. Data will only be accessed by the investigator and the supervisor, and the participant's identity will be anonymised using a coding system.

   Conflict of Interest:
4. There will be no conflict of interest in the study.

ELIGIBILITY:
Inclusion Criteria (care home residents):

* Residents' Age: 65 years of age and older living in a care home, and
* Have no cognitive impairment or in case of cognitive impairment have a score of more than 14 on the Montreal Cognitive Assessment (MOCA) screening (Nasreddine et al 2005) and who are able to provide consent or have next-of-kin/relatives/ friends who can give consent on their behalf.

Inclusion criteria (care home employee):

• All full time care home employees and part-time employees who work in the care home on a long-term basis and interact with the care home residents

Exclusion criteria (care home residents):

* 65 years of age and above residents who score less than 14 on the MOCA screening will have moderate to severe cognitive impairment as they may not be able to follow the intervention and tests, or
* with physical or neurological condition that impedes the usage of the hand grip dynamometer, or
* with skin contraindications to wearing an accelerometer, or
* Known to have a diagnosis of severe dementia or other health conditions that contraindicate their participation in the study, or
* residents with cognitive impairment where English is not primary language as screening test is language sensitive, or
* residents who are registered blind with or without mild cognitive impairment

Exclusion criteria (care home employees):

• Part time employees who work on an ad hoc basis and only have intermittent/minimal interaction with care home residents

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Accelerometer(Actigraph) | Pre-intervention for 7 days
  To measure the level of physical activity
Accelerometer(Actigraph) | 3 months post-intervention
  To measure the level of physical activity
Accelerometer(Actigraph) | 6 months post-intervention
  To measure the level of physical activity
Barthel Index | Pre-intervention
  To measure the independence in performing activities of daily living
Barthel Index | 3 months post-intervention
  To measure the independence in performing activities of daily living
Barthel Index | 6 months post-intervention
  To measure the independence in performing activities of daily living
Hand grip dynamometer | Pre-intervention
  To measure their grip strength by using their hands to grip the dynamometer
Hand grip dynamometer | 3 months post-intervention
  To measure their grip strength by using their hands to grip the dynamometer
Hand grip dynamometer | 6 months post-intervention
  To measure their grip strength by using their hands to grip the dynamometer
Simplified Nutritional Appetite Questionnaire (SNAQ) | Completed pre-intervention
  Self-administered questionnaire that will measure appetite levels
Simplified Nutritional Appetite Questionnaire (SNAQ) | Completed 3 months post-intervention and 6 months post intervention
  Self-administered questionnaire that will measure appetite levels
Simplified Nutritional Appetite Questionnaire (SNAQ) | Completed 6 months post-intervention
  Self-administered questionnaire that will measure appetite levels
EQ-5D-5L questionnaire | Completed pre-intervention
  self-administered questionnaire that will measure quality of life
EQ-5D-5L questionnaire | Completed 3 months post-intervention and 6 months post intervention
  self-administered questionnaire that will measure quality of life
EQ-5D-5L questionnaire | Completed 6 months post-intervention
  self-administered questionnaire that will measure quality of life
Focus group discussion for care home staff | Conducted at the 6 month timeline of data collection
  this will be a guided discussion facilitated by the researcher to understand the feasibility of implementing personalised interactive exercises & activities in a care home

CONTACTS AND LOCATIONS:
Overall Officials: Jane Murphy, Study Director — Professor of Nutrition

IPD SHARING:
Plan to Share IPD: No
Individual participant data are strictly confidential and will not be accessed by researcher. This will be assessed by care home staff.

REFERENCES:
- [Background] Bradshaw SA, Playford ED, Riazi A. Living well in care homes: a systematic review of qualitative studies. Age Ageing. 2012 Jul;41(4):429-40. doi: 10.1093/ageing/afs069. Epub 2012 Jun 7. PMID 22678747